CLINICAL TRIAL: NCT01391455
Title: Isolation of the Spermatic Cord Following Mesh Inguinal Hernia Repair
Brief Title: Isolation of the Spermatic Cord in Mesh Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chatham Kent Health Alliance (Other)
Responsible Party: John A. Morrison. Chief of Surgery, Chatham Kent Health Alliance
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: mesh isolation
Record Dates: First submitted 2011-07-06; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Inguinal Hernia
Keywords: Inguinal hernia repair; Mesh; Groin pain; Testicular pain
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spermatic Cord in contact with mesh (No Intervention): Where the spermatic cord has been allowed to remain in contact with the mesh.
- Spermatic Cord is isolated from the mesh (Experimental): The inguinal ligament is interposed between the cord and the mesh and then repaired. This isolates the cord from the mesh and the splinting function of the overlying inguinal ligament.
  Interventions: Procedure: Isolation of the spermatic cord from mesh

INTERVENTIONS:
Procedure: Isolation of the spermatic cord from mesh — The spermatic cord is isolated from the mesh employed to repair an inguinal hernia following standard open repair.
  Arms: Spermatic Cord is isolated from the mesh

SUMMARY:
There are in excess of 1 million operations performed annually to repair inguinal hernias, mostly in the male population. Unfortunately, some patients continue to suffer both groin or testicular pain for varying lengths of time postoperatively. This can lead to a severe degradation of the patient's lifestyle, work habits and sexual function. The origin of the pain is felt to be secondary to the inflammatory reaction caused by the mesh. This also involves the spermatic cord and its structures, leading to orchidinia and possibly azospermia.

DETAILED DESCRIPTION:
In this prospective randomized trial, male patients with a primary symptomatic unilateral inguinal hernia will be admitted to the trial. All patients must be over 21 years of age. In order to avoid inguinal nerve entrapment or damage by mesh fixation sutures Covidien Parietene ProGrip mesh will be employed. This mesh does not require fixation. Standard open inguinal hernia repair will take place with nerve preservation, as day surgery cases. In the randomized portion of the study, the mesh will be placed as usual along the posterior wall of the inguinal canal, however the inguinal ligament will be interposed between the mesh and the spermatic cord, thus isolating the cord from intimate contact with the mesh, and a reduction in postoperative inflammatory changes.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a primary unilateral inguinal hernia

Exclusion Criteria:

* Medically unfit for surgical repair

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of groin or testicular pain lasting longer than 3 months postoperatively. | 1 year postoperatively
  All patients will be evaluated using the Carolina's Comfort Scale

SECONDARY OUTCOMES:
Number of patients with adverse events. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John A Morrison, MD;FRCS(C), Principal Investigator — Chatham Kent Health Alliance
Locations (1):
- Chatham Kent Health Alliance, Chatham, Ontario, Canada